CLINICAL TRIAL: NCT04738188
Title: Efficacy and Safety of TACE on Downstaging Hepatocellular Carcinoma Beyond UCSF Criteria: a Multi-center, Randomized, Parallel-controlled Study
Brief Title: Efficacy and Safety of TACE on Downstaging Hepatocellular Carcinoma Beyond UCSF Criteria;
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19229-0-02
Record Dates: First submitted 2020-11-23; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Epirubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-eluting bead transarterial chemoembolization(DEB-TACE) (Experimental)
  Interventions: Procedure: DEB-TACE; Device: Drug-eluting Beads; Drug: Epirubicin
- conventional transarterial chemoembolization(cTACE) (Active Comparator)
  Interventions: Procedure: cTACE; Drug: Epirubicin

INTERVENTIONS:
Procedure: DEB-TACE — Drug-eluting beads transcatheter arterial chemoembolization
  Arms: Drug-eluting bead transarterial chemoembolization(DEB-TACE)
Procedure: cTACE — Transcatheter arterial chemoembolization
  Arms: conventional transarterial chemoembolization(cTACE)
Device: Drug-eluting Beads — Drug-eluting beads
  Arms: Drug-eluting bead transarterial chemoembolization(DEB-TACE)
Drug: Epirubicin — Chemotherapy drug for intra-arterial infusion

SUMMARY:
This is a multicenter, randomized, parallel controlled study to determine the efficacy and safety of transcatheter arterial chemoembolization (TACE) on downstaging hepatocellular carcinoma beyond University of California, San Francisco (UCSF) criteria.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 70 years of age, of any sex;
2. Patients who have histopathological or cytological proof of hepatocellular carcinoma (HCC) or meet the diagnostic criteria of Diagnosis, management, and treatment of hepatocellular carcinoma(V2017);
3. Beyond UCSF criteria: Diameter of single HCC lesion is between 6.5 cm and 10 cm; The number of tumors ≤3 with the maximum diameter of 4.5-5cm and the total diameter ≤10cm; Multiple HCC lesions ≤5 nodules, each lesion diameter≤4 cm with a total diameter ≤10 cm. Patients cannot be treated with resection or liver transplantation;
4. Patients with stage Ib，IIa，IIb in China liver cancer staging (CNLC) ;
5. Child-Pugh's grade A or B (no more than 7 score);
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-1;
7. Patients with hepatitis B virus (HBV) infection should receive routine antiviral therapy;
8. The function of main organs is normal and meet the following criteria:

1) Outcome of blood routine must meet the following criteria (No blood transfusion or blood products were performed within 4 days, and no g-CSF or other hematopoietic stimulants were used for correction): i. Hemoglobin(HB)≥90 g/L; ii. Absolute neutrophil count (ANC)≥1.5×109/L； iii. Platelet (PLT)≥80×109/L; 2) Outcome of hemal biochemistry examination meet the following criteria: i. Albumin (ALB) ≥29 g/L; ii. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)<2.5 × upper limit of normal (ULN); iii. Total bilirubin (TBIL) ≤2 × ULN; iv. Serum creatinine (SCr) ≤1.25 × ULN, or endogenous creatinine clearance > 45 ml/min (Cockcroft-Gault formula); 3) Patients who have normal livers with an Remnant Liver Volume (RLV)/Standard Liver Volume(SLV) >20% ; Patients who have cirrhosis with an RLV/SLV>40%; 9. Life expectancy of > 3 months; 10. Patients volunteered to participate in this study and signed informed consent, with good compliance.Exclusion Criteria.

Exclusion Criteria:

1. Patients with extrahepatic metastasis or main portal vein /main hepatic vein invasion;
2. Patients with diffuse liver cancer;
3. Patients with myocardial ischemia, myocardial infarction or poor controlled arrhythmia (including QTc≥470 ms) beyond stage Ⅱ; according to New York Heart Association (NYHA) standard, patients with heart failure in stage Ⅲ～Ⅳ; patients with an left ventricular ejection fraction(LVEF) <50%;
4. Abnormal coagulation （International Normalized Ratio(INR)>1.5, Prothrombin Time(PT)>ULN+4s or Activated Partial Thromboplastin Time (APTT) >1.5 ×ULN）,or patients with bleeding tendency or undergoing thrombolytic or anticoagulant therapy;
5. Patients unsuitable for the study in the opinion of the Investigator;
6. Pregnant or breastfeeding women; women of childbearing ages unless using effective contraception;
7. Patients with mental disorders or history of abuse of psychotropic substances;
8. Infection with human immunodeficiency virus (HIV);
9. A history of liver resection, liver transplantation, interventional therapy, or combined with other malignant tumors;
10. Patients with active infection;
11. Patients with contraindications to TACE or epirubicin;
12. Floating population or with poor compliance;
13. Patients in other clinical trials conducting with experimental-related drugs or devices within 4 weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2020-03-18 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Downstaging success rate | Within 6 months after surgery
  Criteria for success rate in downstaging meet UCSF criteria or the standard for liver resection.

SECONDARY OUTCOMES:
Complete response (CR) | 1, 3, 6 months after surgery
  Disappearance of any intratumoral arterial enhancement in all target lesions
Partial response (PR) | 1, 3, 6 months after surgery
  At least a 30% decrease in the sum of diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions
Stable disease (SD) | up to 6months after TACE procedure
  Number of the subjects that do not qualify for partial response or progressive disease measured by modified Response Evaluation Criteria in Solid Tumors( mRECIST) criteria
Progressive disease (PD) | 1, 3, 6 months after surgery
  An increase of at least 20% in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since treatment started
Objective response (OR) | 1, 3, 6 months after surgery
  CR+PR
Duration of downstaging | within 36 months
  Interval between initial TACE treatment and the success or failure of downstaging according to the UCSF criteria assessed by the dynamic enhanced CT ;
Times of TACE treatments | within 36 months
  Times of TACE surgery
Changes of tumor biomarkers (AFP, PIVKA-Ⅱ) | From 7 days before TACE or curative treatments to the endpoints of the trial.(Up to 36 months)
  AFP and PIVKA-II must be measured at 1week before, 1 week,1month after TACE or curative treatment; AFP ,PIVKA-II could be measured every 3-6 months during follow up according to the availability of equipment at the site
Changes in liver function | from the date of the first TACE to the end of the clinical trial or the death of the patient，Up to 36months
  Changes of the Child-pugh Score that used to assess the prognosis of chronic liver disease,consisting of 5 items(ascites,total bilirubin，albumin,prothrombin time and degree of encephalopathy),of which is scored 1-3 points,with 3 indicating greatest severity)
Tumor-free survival (TFS) | Within 36 months
  as the time from surgery initiation to tumor recurrence or death from any cause
Progression-free survival (PFS) | Within 36 months
  as the time from surgery initiation to disease progression or death from any cause
Overall survival (OS) | Within 36 months
  as the time from surgery initiation to death from any cause
Recurrence rate of Hepatocellular carcinoma | Within 36 months
  Recurrence rate of hepatocellular carcinoma

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No